CLINICAL TRIAL: NCT02018926
Title: A Phase I/II, Multi-Center Study of Mocetinostat (MGCD0103) in Combination With Azacitidine in Subjects With Intermediate or High Risk Myelodysplastic Syndrome (MDS)
Brief Title: Safety Study of Mocetinostat in Combination With Azacitidine in Subjects With MDS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0103-014
Record Dates: First submitted 2013-12-12; First posted 2013-12-23 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Myelodysplastic Syndrome
Keywords: Mocetinostat; Azacitidine; Vidaza; Myelodysplastic syndrome; HDAC; HMA; MDS
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — mocetinostat; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mocetinostat and azacitidine (Experimental): Drug: Mocetinostat (MGCD0103) Mocetinostat (a histone deacetylase [HDAC] inhibitor) 70 mg or 90 mg dose, oral capsules 3 times weekly beginning on day 5 for 10 doses in each 28 day cycle
  Drug: Azacitidine (Vidaza) Azacitidine (a hypomethylating agent [HMA]) 75 mg/m2 dose, by intravenous (IV) infusion or subcutaneous (SC) injection beginning on day 1 for 7 doses in each 28 day cycle
  Interventions: Drug: Mocetinostat; Drug: Azacitidine

INTERVENTIONS:
Drug: Mocetinostat — Mocetinostat (a histone deacetylase [HDAC] inhibitor) 70 mg or 90 mg dose, oral capsules 3 times weekly beginning on day 5, for 10 doses in each 28 day cycle
  Other Names: MGCD0103
Drug: Azacitidine — Azacitidine (a hypomethylating agent [HMA]) 75 mg/m2 dose, by intravenous (IV) infusion or subcutaneous (SC) injection beginning on day 1 for 7 doses in each 28 day cycle
  Other Names: Vidaza

SUMMARY:
Mocetinostat is an orally administered histone deacetylase (HDAC) inhibitor. Azacitidine is a hypomethylating agent (HMA) used to treat MDS. In this study, patients with intermediate- or high-risk MDS will receive treatment with mocetinostat and azacitidine to evaluate the safety of the study treatment. Safety assessments will include echocardiograms, electrocardiograms and routine safety laboratory studies (hematology and serum chemistry). In addition, clinical response to treatment will be monitored using bone marrow aspirates or biopsies, and other routine methods.

DETAILED DESCRIPTION:
The study will include multiple cohorts of patients. In the first cohort, patients may have previously received treatment with hypomethylating agents such as azacitidine. In later cohorts, prior treatment with this class of anti-cancer agents will be excluded. Later cohorts will include patients that are receiving this class of agents, specifically azacitidine, for the first time.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of intermediate- or high-risk (IPSS criteria) myelodysplastic syndrome.

Cohort 1: Any prior treatment, enrollment complete. Cohort 2: Limited or no prior treatment for MDS. Prior treatment should not include hypomethylating agents such as azacitidine or decitabine, or HDAC inhibitors.

ECOG Performance Status 0 or 1.

Exclusion Criteria:

Current or history of small, moderate or large pericardial effusion, tamponade and/or pericarditis.

Significant cardiac abnormalities such as recent myocardial infarction, congestive heart failure ≥ Class 3, or symptomatic, uncontrolled atrial fibrillation, atrial flutter or sinus tachycardia.

Prolonged QT/QTc interval.

Other active cancer excluding basal cell carcinoma or cervical intraepithelial neoplasia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events, including pericardial events, as a measure of safety | 6 months

SECONDARY OUTCOMES:
Number of subjects experiencing clinical disease response | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Isan Chen, MD, Study Director — Mirati Therapeutics Inc.
Locations (10):
- United States (10):
  - Georegetown University, Washington D.C., District of Columbia
  - Lakes Research, Miami Lakes, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Norris Cotton Cancer Center, Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - New York Medical College, Valhalla, New York
  - Duke University Medical Center, Durham, North Carolina
  - St. Francis Hospital, Greenville, South Carolina
  - Cancer Care Centers of South Texas, New Braunfels, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Fletcher Allen Health Care and Vermont Cancer Center, Burlington, Vermont